CLINICAL TRIAL: NCT01354028
Title: Effects of Massage Therapy to Induce Sleep in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 130342
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-04

CONDITIONS: Premature Birth of Newborn
Keywords: premature infant; massage therapy; sleep induction; relaxation
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Massage therapy (Experimental): Massage therapy for 10 minutes during quiet alert state following 9 AM feeding. Actigraph in place to measure sleep for 3 hours.
  Interventions: Other: Massage therapy
- No massage therapy (No Intervention): This was a crossover trial with two arms. On one day, infants received massage therapy for 10 minutes. On the other day, infants were monitored as usual with the Actigraph to measure sleep efficiency, but received no massage therapy. This was the control or no intervention arm.

INTERVENTIONS:
Other: Massage therapy — An overall massage time of approximately 10 minutes, administered by physical therapists. Almond oil or baby lotion that is currently used in standard care in the ACH NICU will be used to assist with ease of skin to skin contact during moderate pressure massage. Infants will receive two repetitions of 5-1minute periods of 12 strokes lasting approximately 5 seconds each described in protocol. Actigraph device is on infant's ankle to measure sleep.
  Arms: Massage therapy

SUMMARY:
Premature infants sometimes require sedation to ensure minimal movement during diagnostic procedures such as MRIs. However, sedatives may produce adverse effects. The purpose of this two-day study is to determine whether massage therapy will promote sleep in preterm infants and also help them to stay asleep, providing a safer way to sedate infants for procedures. A small instrument called a sleep watch or actigraph will be placed around the infant's ankle to measure muscle activity and provide an indication of sleep. Infants will receive a 10- minute massage on one morning of the study and no massage on the alternate morning. Recordings from the actigraph will show whether there is difference in sleep pattern with and without massage. Infants will be monitored for any heart rate and oxygen saturation changes on both mornings of the study.

DETAILED DESCRIPTION:
This cross-over trial pilot study will assess the effectiveness of massage therapy for inducing and maintaining sleep in preterm infants. Massage therapy promotes relaxation and lowers stress levels, evidenced by increased vagal activity and lower cortisol levels. Safer methods of inducing sleep without drugs would be beneficial for infants who require sedation for diagnostic studies. The sample will include infants over 3 days old and between 32-40 weeks adjusted gestational age in a Neonatal Intensive Care Unit (NICU). Infants who are clinically unstable, require surgery, have major congenital anomalies or have a history of severe birth asphyxia will be excluded.

After parental consent, infants will be randomized to receive massage on study day 1 or study day 2. Standard care will be provided on the alternate study day. A minimum of 30 infants is required to complete the study. The primary outcome measure used to document the response to massage will measured by the Motionlogger® Micro Sleep Watch® Actigraph (Actigraph). The actigraph will be placed on the infant's ankle approximately following the 9 am feed and will record lower extremity activity until approximately the 12 pm feed. Massages will occur after a minimum of 30 minutes following the morning feeding when the infant is in a quiet alert state and will be approximately 10 minutes in length. Baby lotion used as standard care in the NICU will be used to facilitate ease of massage.

Primary outcome measures will include data recorded by the actigraph: (a) sleep onset following massage intervention, (b) sleep end time, (c) number of awakenings and duration of awakenings during the study interval, (d) the duration of the longest sustained sleep period, and (e) sleep efficiency. Secondary outcomes will include oxygen saturation and heart rate during massage and for 30 minutes after massage.

ELIGIBILITY:
Inclusion Criteria

* > 3 days old
* 32-48 weeks adjusted gestational age
* Minimum of 28 weeks gestational age at birth
* Clinically stable as determined by an neonatologist
* Stable respiratory status on room air or nasal cannula flow <2 LPM
* Not meeting exclusion criteria

Exclusion Criteria:

* Documented maternal opiate use prior to admission to Labor and Delivery (opiates administered by physicians' order during labor prior to delivery do not mandate exclusion from the study as long as the mother does not have a past history of opiate abuse or a positive drug screen at hospital admission prior to delivery).
* Clinically unstable and/or unable to be moved from the infant warmer
* Severe congenital anomalies likely to be associated with developmental delay
* Apgar score of ≤ 3 at 5 minutes of age
* Any other condition that in the opinion of the investigator might result in unnecessary or excessive risk to the subject
* Unstable respiratory status
* Sedation in the previous 24 hours before the infant's trial.
* Neurological disease: grade III or IV intraventricular hemorrhage, periventricular leukomalacia, evidence of hypoxic ischemic encephalopathy
* Anticipated painful procedures during the study period between 9 am and 12 pm

Ages: 3 Days to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Hall, M.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants were recruited from the Neonatal Intensive Care Unit (NICU) at a Children's Hospital. Recruitment dates were 03/09/2011 to 05/09/2012. A total of 30 infants were enrolled.
Pre-assignment Details: Seven infants were enrolled but did not complete the study. Two infants developed medical complications before the study and therefore became ineligible. Four infants were discharged before the study began. One infant did not have a quiet alert state after feeding and the study was discontinued at that point with no data collected.
Groups:
- Massage Therapy First Day, no Massage Therapy Second Day: Day one of study: Massage therapy for 10 minutes during quiet alert state following 9 AM feeding. Actigraph in place to measure sleep for 3 hours.
  Day two of study: No massage therapy. Actigraph in place to measure sleep for 3 hours
- No Massage Therapy First Day, Massage Therapy Second Day: Day one of study: No massage therapy. Actigraph in place to measure sleep for 3 hours.
  Day two of study: Massage therapy for 10 minutes during quiet alert state following 9 AM feeding. Actigraph in place to measure sleep for 3 hours.
Period: Overall Study
Arm/Group | Massage Therapy First Day, no Massage Therapy Second Day | No Massage Therapy First Day, Massage Therapy Second Day
Started | 15 | 15
Completed | 13 | 10
Not Completed | 2 | 5
Not completed — Physician Decision | 0 | 2
Not completed — Discharged before study start | 2 | 2
Not completed — No quiet alert state | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Massage Therapy
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  newborn infant >3 days | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Quality of Sleep, Defined by Number and Duration of Awakenings, and Longest Sustained Sleep Period for the Study Interval. These Data Were Measured by the Actigraph Software and Summarized as Percentage of Time Spent Sleeping, or Sleep Efficiency
Description: Sleep onset following the first quiet alert state after the 9 AM feed Sleep end time Number of awakenings and duration of the awakenings during the study period Longest sustained sleep period for the study interval Percentage of time spent sleeping, or sleep efficiency, will be used to summarize the data, comparing sleep efficiency over 2 days and using each infant as his/her own control
Time Frame: Participants were followed for two days
Population: A convenient number of participants was selected for this pilot study.
Measure: Mean (Standard Deviation); unit: percentage of time spent sleeping
Groups:
- Sleep Efficiency With Massage Therapy: Massage therapy for 10 minutes during quiet alert state following 9 AM feeding. Actigraph in place to measure sleep efficiency for 3 hours - following 9 AM feeding until approximately 12 noon.
- Sleep Efficiency With no Massage Therapy: No intervention. This is a crossover trial. Infants received massage therapy on one day and no massage (no intervention) on the other day. They continued to be monitored for sleep efficiency using the Actigraph on the day that they received no intervention, but at corresponding times. Actigraph in place to measure sleep efficiency for 3 hours - following 9 AM feeding until approximately 12 noon.
Arm/Group | Sleep Efficiency With Massage Therapy | Sleep Efficiency With no Massage Therapy
Number analyzed (Participants) | 23 | 23
percentage of time spent sleeping | 78.7 (20) [-3.5 to 12.9] | 77.8 (21.4)
Statistical Analysis 1: Comparison: Sleep Efficiency With Massage Therapy vs Sleep Efficiency With no Massage Therapy; Null hypothesis: there will be no difference in sleep efficiency in preterm infants on the day of massage versus the day without massage. Power calculation: the sample size was determined by convenience for this pilot study; Test type: Superiority or Other; p = 0.1303, Chi-squared; Degrees of freedom =1

2. Secondary Outcome: Oxygen Saturation Levels During Massage
Description: Infants in the NICU are routinely attached to pulse oximeter monitors that measure oxygen saturation continuously. If the infant is stressed, oxygen levels may drop. Oxygen saturation was monitored during massage therapy as a routine measure but also to ensure that infants did not become stressed during the massage.
Time Frame: During massage
Population: We determined a convenient size for this pilot study
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- Oxygen Saturation During Massage: Oxygen saturation during massage therapy
- Oxygen Saturation Without Massage: No intervention. This is a crossover trial. Infants received massage therapy on one day and no massage (no intervention) on the other day. They continued to be monitored for heart rate, oxygen saturation, and sleep efficiency using the Actigraph on the day that they received no intervention, but at corresponding times.
Arm/Group | Oxygen Saturation During Massage | Oxygen Saturation Without Massage
Number analyzed (Participants) | 23 | 23
percentage of oxygen saturation | 99.7 (0.7) [98 to 99] | 99.3 (1.18)

3. Secondary Outcome: Heart Rate
Description: Heart rate during massage therapy
Time Frame: During massage therapy
Population: A convenient size was determined for this pilot study
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Heart Rate During Massage: Heart rate during massage therapy
- Heart Rate Without Massage: No intervention. This is a crossover trial. Infants received massage therapy on one day and no massage (no intervention) on the other day. They continued to be monitored for heart rate, oxygen saturation, and sleep efficiency using the Actigraph on the day that they received no intervention, but at corresponding times.
Arm/Group | Heart Rate During Massage | Heart Rate Without Massage
Number analyzed (Participants) | 23 | 23
beats per minute | 162.5 (12.7) | 169.45 (12.86)

4. Primary Outcome: Number of Infants Sleeping at the End of the Massage Period
Description: Investigators compared the number of infants sleeping at the end of the massage period with the percentage of infants sleeping at the same time on the non massage day.
Time Frame: Minute massage ended
Population: A convenient number of infants was determined for this pilot study
Measure: Number; unit: participants
Groups:
- No Massage Therapy: This was a crossover trial. The infants received 10 minutes of massage therapy on one day, and no massage therapy (no intervention) the other day. On the day that infants did not receive massage therapy, they were monitored as usual with heart rate and oxygen saturation levels and with the Actigraph that measured sleep efficiency, but there was no intervention.
Arm/Group | Massage Therapy | No Massage Therapy
Number analyzed (Participants) | 23 | 23
participants | 7 | 14
Statistical Analysis 1: Comparison: Massage Therapy vs No Massage Therapy; Null hypothesis: there is no difference in massage therapy or no massage therapy in number of infants who will be asleep at the end of massage or the corresponding time frame on the non massage day. Pearson's chi square=4.98; Test type: Superiority or Other; p = 0.026, Chi-squared — Pearson's chi square; Degrees of freedom=1

ADVERSE EVENTS:
Time Frame: Infants were enrolled in the study three hours per day for two days. They received massage therapy on one day and no massage therapy on the other day (crossover trial). Data were collected for a total period of 1 year, 2 months.
Arm/Group | Massage Therapy | No Massage Therapy
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
The sample size was small. 30 infants were enrolled, but 7 infants were discharged or became ineligible and could not start the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes